CLINICAL TRIAL: NCT01068847
Title: Drug Discrimination in Methadone-Maintained Humans Study 3
Acronym: OMDD3
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Arkansas (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Basic Science
Other Study IDs: R01DA010017-03 (NIH); R01DA010017-03 (NIH); 110528; R01DA010017 (NIH); DPMC (Other: NIDA)
Record Dates: First submitted 2010-02-12; First posted 2010-02-15 (Estimated); Last update posted 2013-03-07 (Estimated); Status verified 2013-03

CONDITIONS: Drug Dependence
Keywords: Opioid dependence; methadone; opioid
MeSH Terms: conditions — Substance-Related Disorders; Opioid-Related Disorders | interventions — Cycloserine; Naloxone; Nifedipine; Sodium Chloride; tizanidine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Receives 2-4 of the drugs listed under Intervention
  Interventions: Drug: 2-4 of the drugs listed below

INTERVENTIONS:
Drug: 2-4 of the drugs listed below — Cycloserine: 500, 675, 750 mg oral capsules may possibly given. Naloxone: 0.15mg/70Kg or 0.2mg/70kg I.M. injection may possibly be given. Nifedipine: 10, 20 mg oral capsules may possibly be given. Placebo (sugar pill or microcrystalline cellulose): oral capsules may be given. Saline: I.M. injection may possibly be given. Tizanidine: 4, 8, 12 mg oral capsules may possibly be given. Verapamil: 30, 60, 120 mg oral capsules may possibly be given.
  Other Names: Cycloserine: Seromycin; Naloxone: Narcan; Nifedipine: Adalat, Procardia; Placebo; Saline; Tizanidine: Zanaflex; Verapamil: Veralan

SUMMARY:
This study involves giving psychoactive drugs intramuscularly (injected into the muscle of the upper arm or the hip) and/or orally, and measuring the participant's ability to tell the difference between one drug and another, as well as measuring the effects of the drugs on mood, physiology (e.g., heart rate, blood pressure, respiration rate) and behavior. Each participant will receive 2-4 of the listed interventions.

ELIGIBILITY:
Inclusion Criteria:

1. Must be between the ages of 18-65.
2. Participation in the UAMS Substance Abuse Treatment Clinic Methadone Maintenance Program or the CATAR Clinic Little Rock with maintenance on a stable dose of methadone (+ or - 10 mg) for at least 1 month prior to study entry.
3. Subjects would have to be in "good standing" in the methadone maintenance program in order to participate; i.e., compliance with scheduled medication and group therapy session hours. This would be defined as < 3 missed methadone medications and missed < 3 group and <3 individual therapy sessions in the two months prior to study participation
4. Subjects must submit a urine sample negative for illicit drugs prior to study entry.
5. Subjects must be able to read and understand English.

Exclusion Criteria:

1. Unstable medical condition (e.g., major, unstable cardiovascular, renal, endocrine or hepatic disease) or stable medical condition requiring treatment that would interact with study medications (e.g., controlled hypertension on an antihypertensive) or ability to participate in study sessions, (e.g.,chronic back pain that would preclude being able to sit for long periods, etc), to be determined by history provided by the prospective subject or laboratory evaluation and physical examination as outlined below. These would be determined by the study physician alone or in consultation with the PI.
2. Current diagnosis of other drug or alcohol physical dependence (other than tobacco).
3. History of major psychiatric disorder (psychosis, schizophrenia, bipolar) or current psychiatric disorder that requires medication (e.g., current major depression).
4. Pregnancy, plans to become pregnant or inadequate birth control (adequate birth control includes an IUD, condoms, birth control pills, etc). Male participants are encouraged to use condoms because little has been studied on the effects of these drugs on the male reproductive system.
5. Present or recent use of over-the-counter psychoactive drug, prescription psychoactive drug (antidepressants, anxiolytics, antipsychotics and anticonvulsants that may also be used for mood stabilization or sleep disruption) or drug (e.g., ciprofloxacin, fluvoxamine) that would have major interaction with drugs to be tested.
6. Liver function tests greater than 3 times normal, BUN and Creatinine outside normal range, or thyroid function tests outside normal range.
7. A supine or semi-recumbent blood pressure of 100/65mmHg, a seated blood pressure of 90/60mmHg, or orthostatic change of >20mmHg systolic or >10mmHg diastolic on standing or heart rate less than 60 beats/min.
8. EKG abnormalities including but not limited to: bradycardia (<60 bpm); prolonged QTc interval (>450 msec); Wolff-Parkinson White syndrome; wide complex tachycardia; 2nd degree, Mobitz type II heart block; 3rd degree heart block; left or right bundle branch block.
9. Participants who become arrested and/or incarcerated will not be allowed to continue to participate.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2010-02; Primary Completion 2012-10 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Drug Discrimination Performance | Every Session

SECONDARY OUTCOMES:
Self-Report Ratings | Every Session
Vital Signs | Every session
ECG | Test Sessions

CONTACTS AND LOCATIONS:
Overall Officials: Alison Oliveto, Ph.D., Principal Investigator — University of Arkansas
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States